CLINICAL TRIAL: NCT01565993
Title: Is the Use of Prophylactic Hemoclips in the Endoscopic Resection of Large Pedunculated Polyps Useful? A Prospective and Randomized Study
Brief Title: The Use of Prophylactic Hemoclips in the Endoscopic Resection of Large Pedunculated Polyps
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The unexpected increase in morbidity of the hemoclip group
Sponsor: Hospital Severo Ochoa (Other)
Responsible Party: Principal Investigator, Elvira Quintanilla, Physician, Hospital Severo Ochoa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EQCLIPS
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Results first posted 2012-05-25 (Estimated); Last update posted 2012-05-25 (Estimated); Status verified 2012-04

CONDITIONS: Postpolypectomy Bleeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hemoclip (Active Comparator): In group HEMOCLIP, one or more clips were placed (based on the criteria of the endoscopist in accordance with the size of the pedicle), and the polyp was subsequently resected using a diathermy loop
  Interventions: Device: Hemoclip
- Conventional Polipectomy (Active Comparator): In group CONVENTIONAL POLYPECTOMY, a conventional polypectomy was performed, which was not aided beforehand by any other hemostatic technique
  Interventions: Device: Conventional Polipectomy

INTERVENTIONS:
Device: Hemoclip — A rotatable clip-fixing device "Quickclip 2" standard was used (Olympus Medical Systems Corp. Hachioji-shi, Tokyo, Japan), with an opening diameter of 135º and a maximum insertion portion diameter of 2.6 mm
  Arms: Hemoclip
Device: Conventional Polipectomy — Disposable electrosurgical snares (Olympus Medical Systems Corp. Hachioji-shi, Tokyo, Japan) and an electrosurgery unit ERBE (ERBE Elektromedizin GmbH, Germany) were used for polyp resection
  Arms: Conventional Polipectomy

SUMMARY:
The aim of our study is to analyze the advantages of the prophylactic use of hemoclips before polypectomy in our usual clinical practice, through a prospective randomized study that determines their effectiveness compared to conventional polypectomy, assessing the decrease in immediate and delayed post-polypectomy bleeding

DETAILED DESCRIPTION:
The methods for preventing post-polypectomy bleeding (PPB) are not standardised and there are groups that use hemoclips for this purpose.

The aim of our study is to analyze whether the use of hemoclips reduces PPB complications. It is a prospective, randomised study of patients with pedunculated polyps larger than 10mm. The patients were included in two groups (hemoclip before polypectomy -HC- and standard polypectomy -SP-)

ELIGIBILITY:
Inclusion Criteria:

* Patients with one or more pedunculated polyps, the heads of which measured more than 1cm (regardless of the stalk thickness and length), and they were compared against the size of the biopsy forceps (6mm) and subsequently confirmed in the anatomical specimen
* Not to have any hemostatic alterations at the time the endoscopy was performed (confirmed by the usual blood tests taken before the procedure).

Exclusion Criteria:

* Patients younger than 18 years of age
* Patients with a platelet count of less than 50000, INR larger than 1.5
* Patients who refused to give their informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2007-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elvira M Quintanilla, MD, Principal Investigator — Hospital Universitario Severo Ochoa; Luis R Rábago, PhD, Study Director — Hospital Universitario Severo Ochoa
Locations (1):
- Hospital Universitario Severo Ochoa, Leganés, Madrid, Spain

REFERENCES:
- [Derived] Quintanilla E, Castro JL, Rabago LR, Chico I, Olivares A, Ortega A, Vicente C, Carbo J, Gea F. Is the use of prophylactic hemoclips in the endoscopic resection of large pedunculated polyps useful? A prospective and randomized study. J Interv Gastroenterol. 2012 Oct;2(4):183-188. doi: 10.4161/jig.23741. Epub 2012 Oct 1. PMID 23687606
- [Derived] Quintanilla E, Castro JL, Rabago LR, Chico I, Olivares A, Ortega A, Vicente C, Carbo J, Gea F. Is the use of prophylactic hemoclips in the endoscopic resection of large pedunculated polyps useful? A prospective and randomized study. J Interv Gastroenterol. 2012 Apr;2(2):99-104. doi: 10.4161/jig.22210. Epub 2012 Apr 1. PMID 23687598

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 2007 to 2010, the patients were selected at the digestive endoscopy unit.All of the consecutive patients referred for colonoscopy to the endoscopy office were informed of the aims of the ongoing research and were invited to take part in the study for which they gave their informed consent before the endoscopic procedure was performed
Pre-assignment Details: Where more than one polyp was observed in a patient, all the polyps were included in the same randomization group, so that they all underwent the same technique (conventional or modified polypectomy). 3 patients were excluded for failing to meet the inclusion criteria since they involved semi-pedunculated polyps measuring less than 1cm.
Groups:
- Group A: Hemoclips: In group A, one or more clips were placed (based on the criteria of the endoscopist in accordance with the size of the pedicle), and the polyp was subsequently resected using a diathermy loop
- Group B: Conventional Polipectomy: In group B, a conventional polypectomy was performed, which was not aided beforehand by any other hemostatic technique
Period: Overall Study
Arm/Group | Group A: Hemoclips | Group B: Conventional Polipectomy
Started | 66 | 42 (3 patients were excluded for failing to meet the inclusion criteria)
Completed | 66 (A total of 105 polypectomies were performed on 98 patients) | 39
Not Completed | 0 | 3
Not completed — Physician Decision | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: Hemoclips | Group B: Conventional Polipectomy | Total
Number analyzed (Participants) | 66 | 42 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 65 | 41 | 106
  >=65 years | 1 | 1 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 64.05 (10.99) | 65.55 (12.68) | 64.5 (11.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 49 | 24 | 73
Region of Enrollment [Number; unit: participants]
  Spain | 66 | 42 | 108

OUTCOME MEASURES:

1. Primary Outcome: The Number of Polyps With Complications After Polypectomy (The Total Complication Rate)
Description: In order to test the ability of prophylactic hemoclipping to prevent post-polypectomy bleeding, the investigators were required to register all the adverse events that occurred. These adverse events were called "complications", despite their severity and clinical significance
Time Frame: Between four and six weeks after the polypectomy, the patients were contacted by phone in order to confirm the absence of delayed bleeding
Population: Based on an anticipated decrease of at least 12% in the rate of adverse bleeding events between the group A and the group B, there was an alpha error of 0.05 and a statistical power of 80% with a patient inclusion rate of 1:1. The number of polyps required is 146 per group. Using the Fleiss correction, the final number is 164 per group.
Measure: Number; unit: polyps
Units Other Than Participants: Polyps
Groups:
- Hemoclip: In group HEMOCLIP, one or more clips were placed (based on the criteria of the endoscopist in accordance with the size of the pedicle), and the polyp was subsequently resected using a diathermy loop. In all the polypectomies that were assigned to group HEMOCLIP, a rotatable clip-fixing device "Quickclip 2" standard was used (Olympus Medical Systems Corp. Hachioji-shi, Tokyo, Japan), with an opening diameter of 135º and a maximum insertion portion diameter of 2.6 mm
- Conventional Polipectomy: In group CONVENTIONAL POLYPECTOMY, a conventional polypectomy was performed, which was not aided beforehand by any other hemostatic technique.Disposable electrosurgical snares (Olympus Medical Systems Corp. Hachioji-shi, Tokyo, Japan) and an electrosurgery unit ERBE (ERBE Elektromedizin GmbH, Germany) were used for polyp resection.
Arm/Group | Hemoclip | Conventional Polipectomy
Number analyzed (Participants) | 63 | 35
Number analyzed (Polyps) | 66 | 39
polyps | 7 | 3

2. Secondary Outcome: Difficult to Place the Clip
Description: The hemoclips which were incorrectly placed, mainly because the pedicles were very thick and/or short.
Time Frame: During endoscopic procedure was performed (between 2007 and 2010: period over which the study was conducted)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: During the endoscopic procedure
Arm/Group | Group A: Hemoclips | Group B: Conventional Polipectomy
Serious Adverse Events (participants affected / at risk) | 1/66 | 0/39
Other Adverse Events (participants affected / at risk) | 3/66 | 0/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Hemoclips (N=66) | Group B: Conventional Polipectomy (N=39)
Perforation (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Hemoclips (N=66) | Group B: Conventional Polipectomy (N=39)
Mucosal burn (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
Not to reach the sample size established previously in the initial design, implies bias and decreases the strength of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No